CLINICAL TRIAL: NCT02308462
Title: Implementation and Evaluation of a Family-based Intervention Program for Children and Adolescents of Mentally Ill Parents - a Randomized Controlled Multicenter Trial
Brief Title: Implementation and Evaluation of a Family-based Intervention Program for Children of Mentally Ill Parents
Acronym: CHIMPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silke Wiegand-Grefe, Prof. Dr. (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University of Ulm (Other); Universitätsklinikum Leipzig (Other); LWL-Klinikum Gütersloh (Unknown); Vitos Klinik Rheinhöhe (Unknown); Charite University, Berlin, Germany (Other); Cantonal Hospital Winterthur, Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Silke Wiegand-Grefe, Prof. Dr., Professor of clinical psychology, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O1GY1337; U1111-1162-2635 (Other: World Health Organization (Universal Trial Number)); DRKS00006806 (Registry Identifier: German Clinical Trials Register (DRKS))
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Mood Disorders; Neurotic Disorders; Personality Disorders; Substance-Related Disorders
Keywords: children of mentally ill parents; family intervention; randomized controlled trial
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Mood Disorders; Neurotic Disorders; Personality Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHIMPs intervention (Experimental): Family-Intervention
  Interventions: Behavioral: CHIMPS intervention
- Control (No Intervention): The long-term effectiveness of the CHIMPs intervention under conditions of practice will be examined in comparison to a control condition receiving the usual after care (Treatment as usual = TAU); this testing of effectiveness will be performed in due consideration of the health economic aspects.
  The treatment as usual implies that families of the control Group receive the Treatment that is customary in regular care. Thus, these families normally don't receive any post-treatment. If, however, a member of a control group family appears to have an urgent need for treatment (every Family receives a comprehensive diagnostic investigation at the beginning of the study), the respective family will be placed in the ambulatory care system.

INTERVENTIONS:
Behavioral: CHIMPS intervention — CHIMPs intervention (Family-Intervention composed of 8 Topic-related sessions over a period of 6 month, based on the evaluated manual: a preliminary talk with the family, two sessions with the parents, one session with each child, three sessions with the family).
  The sessions are semi-structured and cover the topics illness and coping, education, family relationships and trusting attachement figures, social network and support of the Family. A detailed description of the procedure is found in the Manual (Wiegand-Grefe, Halverscheid & Plass, 2011).
  Arms: CHIMPs intervention

SUMMARY:
In order to identify psychological stress in children and adolescents of mentally ill parents as early as possible, a special intervention program (CHIMPs = Children of mentally ill parents) was developed. The study at hand will implement this intervention program at five sites in Germany and will further evaluate its effectiveness. The CHIMPs intervention is assumed to reduce children's psychopathology and enhance their health related quality of life.

DETAILED DESCRIPTION:
The main purpose of this study is to implement the manualized family intervention CHIMPs (Children of mentally ill parents) for children and adolescents of psychiatrically ill parents aged between 3 and 19 years at the seven participating centres in regular care. The intervention aims at reducing children's psychopathology and enhancing their quality of life in a sustainable way and, moreover, aims at introducing especially remarkable children and adolescents to an early intervention.

The study represents a prospective, randomized and controlled multicenter study (RCT), contrasting one intervention group and one control group (TAU = Treatment as usual) by measurements at baseline and after six, 12 and 18 months. Within the data collection, the perspective of the psychiatrically ill parent, the partner, each child and the therapist will be considered. Children between 3 and 9 years of age will be evaluated only by the parents and the therapist, from 10 years on, an additional self-report form will be filled out by the child. The measurement will be ruled out indirectly (for the pre-post-measurement) as well as directly (at the end of treatment).

For each endpoint, one comprehensive mixed model will be fitted to the data containing the baseline value and further relevant patient characteristics as covariates, the random group as factor and cluster (center, therapy group, family) as random effect. Missing values will be treated by direct imputation to allow an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Family with at least one psychiatrically ill parent and at least one child between the age of 3 and 19 years
* Consent to participate in the study
* Sufficient knowledge of the German language of parents and children

Exclusion Criteria:

* Severe psychiatric disorders and impairments with acute symptoms such as suicidal tendencies, massive self-injurious behaviour, acute psychotic symptoms etc., making a stationary treatment inevitable and making a ambulatory intervention appear contraindicated (These patients are placed in stationary treatment)
* Children with severe symptoms in the control group will be placed at a participating psychotherapist. Nevertheless, they stay in the control group (as TAU).

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2014-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
children's psychiatric symptomatology (Kiddie-SADS interview) | at the beginning of the study (on study enrolment)
  Children's psychiatric symptomatology will be assessed, in both groups (Intervention group and control group), by an external Independent interview (Kiddie-SADS, Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project (observer-blind rater).
children's psychiatric symptomatology (Child behaviour checklist) | at the beginning of the study (on study enrolment)
  The psychiatric disorders of the children will further be assessed by the CBCL ("Child behaviour checklist", Achenbach, 1991),
children's psychiatric symptomatology (assessed by Youth Self Report) | at the beginning of the study (on study enrolment)
  The psychiatric disorders of the children will further be assessed by the YSR ("Youth self Report", Achenbach, 1991)
children's psychiatric symptomatology (assessed by the SGKJ) | at the beginning of the study (on study enrolment)
  The psychiatric disorders of the children will further be assessed by the SGKJ ("Skala zur Gesamtbeurteilung von Kindern und Jugendlichen", a scale for the overall assessment of children and adolescents, Steinhausen, 1985).
children's psychiatric symptomatology (Kiddie-SADS interview) | after the treatment (after 6 months)
  Children's psychiatric symptomatology will be assessed, in both groups (Intervention group and control group), by an external Independent interview (Kiddie-SADS, Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project (observer-blind rater).
children's psychiatric symptomatology (Kiddie-SADS interview) | after the follow-up period (after 18 months)
  Children's psychiatric symptomatology will be assessed, in both groups (Intervention group and control group), by an external Independent interview (Kiddie-SADS, Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project (observer-blind rater).
children's psychiatric symptomatology (Child behaviour checklist) | after the treatment (after 6 months)
  The psychiatric disorders of the children will further be assessed by the CBCL ("Child behaviour checklist", Achenbach, 1991),
children's psychiatric symptomatology (Child behaviour checklist) | after the follow-up period (after 18 months)
  The psychiatric disorders of the children will further be assessed by the CBCL ("Child behaviour checklist", Achenbach, 1991),
children's psychiatric symptomatology (assessed by Youth Self Report) | after the treatment (after 6 months)
  The psychiatric disorders of the children will further be assessed by the YSR ("Youth self Report", Achenbach, 1991)
children's psychiatric symptomatology (assessed by Youth Self Report) | after the follow-up period (after 18 months)
  The psychiatric disorders of the children will further be assessed by the YSR ("Youth self Report", Achenbach, 1991)
children's psychiatric symptomatology (assessed by the SGKJ) | after the treatment (after 6 months)
  The psychiatric disorders of the children will further be assessed by the SGKJ ("Skala zur Gesamtbeurteilung von Kindern und Jugendlichen", a scale for the overall assessment of children and adolescents, Steinhausen, 1985).
children's psychiatric symptomatology (assessed by the SGKJ) | after the follow-up period (after 18 months)
  The psychiatric disorders of the children will further be assessed by the SGKJ ("Skala zur Gesamtbeurteilung von Kindern und Jugendlichen", a scale for the overall assessment of children and adolescents, Steinhausen, 1985).

SECONDARY OUTCOMES:
children's health related quality of life (Kidscreen) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Kidscreen (Ravens-Sieberer et al., 2006)
parents' health related quality of life (EQ-5D) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  EQ-5D (Brooks, Rabon & de Charro, 2003; Hinz, Klaiberg, Brähler & König, 2006)
Symptomatology of the parents (Brief Symptom Inventory) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Brief Symptom Inventory (Franke, 2000)
Symptomatology of the parents (only Intervention group) (SKID; a structured clinical interview for DSM-IV) | during CHIMPs intervention
  Strukturiertes Klinisches Interview für DSM-IV (SKID; a structured clinical interview for DSM-IV, Wittchen, Zaudig & Fydrich, 1997)
parents' coping with the disorder (Freiburger Fragebogen zur Krankheitsbewältigung) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Freiburger Fragebogen zur Krankheitsbewältigung (FKV; Muthny, 1989)
family relations (children and parents) (Allgemeiner Familienfragebogen) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Allgemeiner Familienfragebogen (FB-A;Cierpka & Frevert, 1995)
Social Support (Oslo Social Support Questionnaire) | at the beginning (on study enrolment) and at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Oslo Social Support Questionnaire (OSSQ; Dalgaard, 1996)
Objectives of the treatment (children and parents) | at the beginning of the study (on study enrolment)
  Objective of the treatment, assessed by the item "What could be the main objective of a possible treatment?"
achievement of the objectives of the treatment (children and parents) | at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  achievement of the objectives of the treatment, assessed by the item "Did you achieve the main objective of your treatment?" and by the item "Taken as a whole, did the family sessions help you?"
Evaluation of the Treatment (children and parents) (Fragebogen zur Beurteilung der Behandlung) | at the end of the intervention (after 6 months) as well as after the follow-up period (after 18 months)
  Fragebogen zur Beurteilung der Behandlung (FBB; Mattejat & Remschmidt, 1999)
health economic assessment of treatment costs (children) (German version of the "Children and adolescent mental health Services receipt inventory) | at the beginning (on study enrolment), at the end of treatment (after 6 months), after 12 months and after the follow-up period (after 18 months)
  German version of the Children and adolescent mental health Services receipt inventory" (CAMHSRI; Kilian et al., 2009)
health economic assessment of treatment costs (parents) (German version of the Client Socioeconomic and Services Receipt Inventory) | at the beginning (on study enrolment), at the end of treatment (after 6 months), after 12 months and after the follow-up period (after 18 months)
  German version of the "Client Socioeconomic and Services Receipt Inventory" (CSSRI; Roick et al., 2001)
Symptomatology of the parents | at the beginning (on study enrolment)
  German version of the "Patient Health Questionnaire" (PHQ; Löwe, Spitzer, Zipfel & Herzog, 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Silke Wiegand-Grefe, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (14):
- Germany (13):
  - Charité Campus Virchow Klinikum, Klinik für Psychiatrie, Psychosomatik und Psychotherapie des Kindes- und Jugendalters, Berlin
  - Vitos psychiatrische Ambulanz Eltville, Eltville
  - Bezirkskrankenhaus Günzburg, Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Günzburg
  - LWL-Klinikum Gütersloh, Klinik für Allgemeine Psychiatrie und Psychotherapie, Gütersloh
  - Schön Klinik Hamburg Eilbek, Abteilung für Psychiatrie und Psychotherapie, Hamburg
  - University Medical Center Hamburg-Eppendorf, Clinic and Polyclinic for psychiatry and psychotherapy, Hamburg
  - Asklepios Klinikum Harburg, Harburg
  - Vitos psychiatrische Ambulanzen Idstein, Idstein
  - Universitätsklinikum Leipzig, Klinik für Psychiatrie, Psychotherapie und Psychosomatik des Kindes- und Jugendalters, Leipzig
  - Universitätsklinkum Leipzig, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Leipzig
  - LWL-Klinik Paderborn, Allgemeine Psychiatrie und Psychotherapie, Paderborn
  - Klinik für Psychiatrie und Psychotherapie des Sächsischen Krankenhauses Altscherbitz, Schkeuditz
  - Vitos psychiatrische Tageskliniken Wiesbaden, Wiesbaden
- Centre of Social Pediatrics, Dept. of Pediatrics and Adolescent Medicine, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krohn L, Deneke C, Wiegand-Grefe S. [Children of depressive parents and psychiatrically inconspicuous parents in the child and adolescent psychiatry--a comparison study]. Prax Kinderpsychol Kinderpsychiatr. 2008;57(7):536-54. doi: 10.13109/prkk.2008.57.7.536. German. PMID 18924530
- [Background] Pollak E, Bullinger M, Jeske J, Wiegand-Grefe S. [How do mentally ill parents evaluate their children's quality of life? Associations with the parent's illness and family functioning]. Prax Kinderpsychol Kinderpsychiatr. 2008;57(4):301-14. doi: 10.13109/prkk.2008.57.4.301. German. PMID 18575057
- [Background] Pollak E, Wiegand-Grefe S, Hoger D. The Bielefeld attachment questionnaires: overview and empirical results of an alternative approach to assess attachment. Psychother Res. 2008 Mar;18(2):179-90. doi: 10.1080/10503300701376365. PMID 18815965
- [Background] Wiegand-Grefe S, Geers P, Petermann F, Plass A. [Children of mentally ill parents: the impact of parental psychiatric diagnosis, comorbidity, severity and chronicity on the well-being of children]. Fortschr Neurol Psychiatr. 2011 Jan;79(1):32-40. doi: 10.1055/s-0029-1245623. Epub 2010 Nov 18. German. PMID 21089005
- [Background] Jeske J, Bullinger M, Wiegand-Grefe S. Do attachement Patterns of parents with a mental illness have an Impact upon how they view the Quality of life of their children? Vulnerable Children and Youth Studies 6(1): 39-50, 2011.
- [Background] Wiegand-Grefe S, Werkmeister S, Bullinger M, Plass A, Petermann F. [Health-related quality of life and social support of children with mentally ill parents: Effects of a manualized family intervention]. Kindheit und Entwicklung 21 (1): 64-73, 2012.
- [Background] Jeske J, Bullinger M, Plass A, Petermann F, Wiegand-Grefe S. [Risk factor coping with a disease: Associations between coping an health related quality of life of children with a mentally ill parent]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie 57 (3): 207-213, 2009.
- [Background] Jeske J, Bullinger M, Wiegand-Grefe S. [Families with mentally ill parents - Connections between Family functioning and health-related life quality of children]. Familiendynamik 35 (4): 338-347, 2010.
- [Background] Wiegand-Grefe S, Halverscheid S, Geers P, Petermann F, Plass A. [Children of mentally ill parents: The relationship between coping with a parental mental illness and children's mental health]. Zeitschrift für Klinische Psychologie und Psychotherapie 39 (1): 13-23, 2010.
- [Background] Wiegand-Grefe S, Jeske J, Bullinger M, Plass A, Petermann F. [Quality of life of children with psychiatrically ill parents: Relationship between characteristics of parental disorder and health-related quality of life of the children estimated by the parents]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie 58 (4): 315-322, 2010.
- [Background] Wiegand-Grefe S, Cronemeyer B, Plass A, Schulte-Markwort M, Petermann F. [Comparison of mental abnormalities in children of mentally ill parents from different points of view: Effects of a manualized family intervention]. Kindheit und Entwicklung 22 (1): 31-40, 2013.
- [Background] Wiegand-Grefe S, Cronemeyer B, Halverscheid S, Redlich A, Petermann F. [Coping strategies of psychiatrically ill parents and psychological abnormalities of their children through the focus of a manualized family intervention]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie 61 (1): 51-58, 2013.
- [Derived] Waldmann T, Schaible J, Stiawa M, Becker T, Wegscheider K, Adema B, Wiegand-Grefe S, Kilian R. The cost-utility of an intervention for children and adolescents with a parent having a mental illness in the framework of the German health and social care system: a health economic evaluation of a randomized controlled trial. Child Adolesc Psychiatry Ment Health. 2023 Dec 21;17(1):141. doi: 10.1186/s13034-023-00693-w. PMID 38129868
- [Derived] Wiegand-Grefe S, Filter B, Busmann M, Kilian R, Kronmuller KT, Lambert M, Norra C, von Klitzing K, Albermann K, Winter SM, Daubmann A, Wegscheider K, Plass-Christl A. Evaluation of a Family-Based Intervention Program for Children of Mentally Ill Parents: Study Protocol for a Randomized Controlled Multicenter Trial. Front Psychiatry. 2021 Jan 20;11:561790. doi: 10.3389/fpsyt.2020.561790. eCollection 2020. PMID 33551858